CLINICAL TRIAL: NCT02224222
Title: Assessment of Frailty as a Risk Factor for Cardiac and Vascular Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Principal Investigator, Andrea Szekely, Associate professor, Semmelweis University
Other Study IDs: VSZÉK-FRAILTY
Record Dates: First submitted 2014-08-14; First posted 2014-08-25 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Intellectual Frailty of Aging; Cardiovascular Diseases; Myocardial Infarction; Vascular Diseases; Heart; Dysfunction Postoperative, Cardiac Surgery
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients undergoing vascular procedures: Including all non-interventional surgical procedures, excluding varix surgery
- Patients undergoing cardiac procedures: Including all non-interventional surgical procedures, excluding HTX

SUMMARY:
The purpose of this study is to assess the impact of frailty as a multidimensional risk factor on the outcomes of adult cardiac and vascular surgery. For the purpose of defining patient frailty a multimodal questionnaire has been developed including measurement of psychological, socioeconomical, neurological and behavioral aspects. This study also features an investigation of the possible relationship between sudden regional weather changes, individual meteorological susceptibility of the patients and the outcomes of adult cardiac and vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients, 18 years or older, admitted to the hospital for elective cardiac or vascular surgery.

Exclusion Criteria:

* Not willing to participate.
* Pregnant women.
* During active psychiatric hospital care.
* Patients with defined legal incapability or limited capability.
* Congenital or acquired speech impediment and locomotion disability of any kind.
* Non-evaluable patient due to communication problems and insufficient clinical information for the judgement of frailty (CFS).
* Patients admitted solely for elective surgery of the varices of the lower extremities.
* Patients with a transplanted heart.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive evaluable patients, 18 years old or older, admitted to Semmelweis University, Heart and Vascular Center for elective cardiac or vascular surgery.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-07; Primary Completion 2020-04 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Length of hospital and intensive care unit stay. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.

SECONDARY OUTCOMES:
The composite of in-hospital death from any cause. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
Evidence of clinically definite postoperative acute kidney injury and the need for dialysis. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
Evidence of clinically definite postoperative low cardiac output syndrome. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
Evidence of clinically definite postoperative cardiac arrythmias. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
Evidence of clinically definite postoperative SIRS. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
Evidence of clinically definite postoperative acute lung injury and the need for mechanical ventilation. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
Evidence of clinically definite postoperative peripheral vascular insufficiency. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
The need for reoperation due to bleeding. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Székely, MD, PhD, Study Director — Semmelweis University, Department of Anesthesiology and Intensive Therapy; Daniel J Lex, MD, Principal Investigator — Semmelweis University Heart and Vascular Center; Nikoletta Czobor, Principal Investigator — Semmelweis University; Peter Misnyovszki, Principal Investigator — Semmelweis University; Hanna Tihanyi, Principal Investigator — Semmelweis University; Kalatin Fink, MD, Principal Investigator — Semmelweis University; Béla Merkely, MD, PhD, DSc, Study Chair — Semmelweis University; László Entz, MD, PhD, Study Chair — Semmelweis University; Zoltán Szabolcs, MD, PhD, Study Chair — Semmelweis University; János Gál, MD, PhD, Study Chair — Semmelweis University; Erzsébet Paulovich, MD, Study Chair — Semmelweis University; Eniko Holndonner-Kirst, MD, Principal Investigator — Semmelweis University
Locations (1):
- Semmelweis University, Heart and Vascular Center, Budapest, Hungary

REFERENCES:
- [Derived] Toth K, Szabo A, Nagy A, Szabo D, Szecsi B, Eke C, Sandor A, Susanszky E, Holndonner-Kirst E, Merkely B, Gal J, Szekely A. Preoperative nutritional state is associated with mid- and long-term mortality after cardiac surgery. Ann Palliat Med. 2021 Nov;10(11):11333-11347. doi: 10.21037/apm-21-1015. Epub 2021 Sep 29. PMID 34670385
- [Derived] Szabo A, Toth K, Nagy A, Domokos D, Czobor N, Eke C, Sandor A, Merkely B, Susanszky E, Gal J, Szekely A. The effect of cognitive dysfunction on mid- and long-term mortality after vascular surgery. BMC Geriatr. 2021 Jan 13;21(1):46. doi: 10.1186/s12877-020-01994-x. PMID 33441102